CLINICAL TRIAL: NCT02440100
Title: An Investigator-and-subject Blind, Phase 1 Study To Characterize The Safety, Tolerability, Pharmacokinetics, And Pharmacodynamics Of Repeat Doses Of Pf-06648671 In Healthy Adult Subjects And Healthy Elderly Subjects
Brief Title: A Phase 1 Study To Characterize The Safety, Tolerability, PK And PK Of Repeat Doses Of PF-06648671 In Healthy Adults And Healthy Elderly Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Triple | Purpose: Basic Science
Other Study IDs: B7991002; 2015-000926-13 (EudraCT Number)
Record Dates: First submitted 2015-05-07; First posted 2015-05-12 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Adult Subjects and Healthy Elderly Subjects
Keywords: Phase 1; Multiple doses of PF-06648671; safety, tolerability, PK; plasma and CSF abeta; drug interaction
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (9):
- Multiple Doses PF-06648671 (Cohort1) (Experimental): Healthy subjects receive 14-day repeated dose once a day at 4 mg of PF-06648671 or matching placebo
  Interventions: Drug: PF-06648671; Drug: Placebo
- Multiple Doses PF-06648671 (cohort 2) (Experimental): Healthy subject receive 14-day repeated dose once a day at 12 mg of PF-06648671 or matching placebo
  Interventions: Drug: PF-06648671; Drug: Placebo
- Multiple doses PF-06648671 (cohort 3) (Experimental): Healthy subject receive 14-day repeated dose once a day at 40 mg of PF-06648671 or matching placebo and CSF LP is collected at baseline and steady state predose on day 1 and 14
  Interventions: Drug: PF-06648671; Drug: Placebo
- Multiple Doses PF-06648671 (cohort 4) (Experimental): Healthy subject receive 14-day repeated dose once a day at 40 mg of PF-06648671 or matching placebo
  Interventions: Drug: PF-06648671; Drug: Placebo
- Multiple Doses PF-06648671 (cohort 5) (Experimental): Healthy subject receive 14-day repeated dose once a day at 100 mg of PF-06648671 or matching placebo, CSF LP is collected at baseline 72 hours prior to day 1 dosing and at steady-state on Day 15, 24 hours after last dosing on day 14
  Interventions: Drug: PF-06648671; Drug: Placebo
- Multiple Doses in Healthy Elderly (cohort 7) (Experimental): Healthy Elderly subjects receive 14-day repeated dose once a day at MTD PF-06648671 defined in healthy adult subjects (part 1)
  Interventions: Drug: PF-06648671; Drug: Placebo
- Multiple Doses PF-06648671 (cohort 8) (Experimental): Healthy subjects receive 14-day repeated dose once a day at 360 mg of PF-06648671 or matching placebo, CSF LP is collected at baseline 72 hours prior to day 1 dosing and at steady-state on Day 15, 24 hours post last dose
  Interventions: Drug: PF-06648671; Drug: Placebo
- Midazolam DDI (optional cohort 9) (Experimental): Healthy Subjects receive single dose of 2 mg midazolam in period 1 followed by 14 days PF-06648671 once a day and coadministration of PF-06648671 and midazolam 2 mg in period 2 (Optional cohort)
  Interventions: Drug: PF-06648671; Drug: Midazolam
- Multiple Doses PF-06648671 (cohort 6) (Experimental): Healthy subject receive 14-day repeated dose once a day at 200 mg of PF-06648671 or matching placebo, CSF LP is collected at baseline 72 hours prior to day 1 dosing and at steady-state on Day 25, 24 hours after last dosing on day 14
  Interventions: Drug: PF-06648671; Drug: Placebo

INTERVENTIONS:
Drug: PF-06648671 — experimental Pfizer compound which will be dosed as oral suspension, once a day for 14 days
Drug: Midazolam — commercial available oral solution of 2 mg midazolam as CYP3A probe substrate for drug interaction evaluation. Midazolam will be given as single dose with and without co-administration of PF-06648671
  Arms: Midazolam DDI (optional cohort 9)
Drug: Placebo — Matching placebo which will be given as oral suspension, once a day for 14 days
  Arms: Multiple Doses PF-06648671 (Cohort1); Multiple Doses PF-06648671 (cohort 2); Multiple Doses PF-06648671 (cohort 4); Multiple Doses PF-06648671 (cohort 5); Multiple Doses PF-06648671 (cohort 6); Multiple Doses PF-06648671 (cohort 8); Multiple Doses in Healthy Elderly (cohort 7); Multiple doses PF-06648671 (cohort 3)

SUMMARY:
This is an investigator-and-subject blind, phase 1 study to characterize the safety, tolerability, pharmacokinetics and central and peripheral pharmacodynamics of 14-day repeated ascending doses of PF-06648671 once a day in healthy adults (part 1) and repeated doses at the maximum tolerated dose (MTD) defined in part 1 in healthy elderly subjects (part 2). The study also include an optional cohort (part 3) to evaluate the drug interaction between PF-06648671 at MTD and CYP3A probe, midazolam

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for enrollment in the study:

1. For Part 1 and Part 3 specific: Healthy female subjects of non childbearing potential and male subjects who, at the time of screening, are between the ages of 18 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead ECG and clinical laboratory tests).
2. For Part 2 specific: Female subjects of non childbearing potential and male subjects who, at the time of screening, are between the age of 65 and 85 years, inclusive. Subjects must be in good health as determined by the Investigator based on a detailed medical history, full physical examination (including blood pressure and pulse rate measurement), 12 lead ECG and clinical laboratory tests. Subjects with mild, chronic, stable disease eg, controlled hypertension, non insulin dependent diabetes, osteoarthritis may be enrolled if deemed medically prudent by the investigator. Subjects taking daily prescription or non prescription medications for management of acceptable chronic medical conditions must be on a stable dose of these, as defined by non change in dose for the 3 months prior to the first dose of study medication and no planned changes during the conduct of the study.
3. Female subjects of non childbearing potential must meet at least one of the following criteria:

   * Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; status may be confirmed by having a serum follicle stimulating hormone (FSH) level confirming the post menopausal state;
   * Have undergone a documented hysterectomy and/or bilateral oophorectomy;
   * Have medically confirmed ovarian failure. All other female subjects (including females with tubal ligations will be considered to be of childbearing potential.
4. Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
5. For Part 2 specific: the creatinine clearance greater than 60 mL/min using the Cockcroft Gault method.
6. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
7. Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

1. For Part 1 and Part 3 specific: Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing) at the discretion of the investigator.
2. For Part 2 specific: Recent (eg, last 6 months) evidence or history of unstable disease or moderate to severe conditions which would, in the Investigator's opinion, interfere with the study evaluations or impact on the safety of participating subjects including but not limited to anemia, liver disease, stroke.
3. Any condition possibly affecting drug absorption (eg, gastrectomy).
4. A positive urine drug screen.
5. History of regular alcohol consumption exceeding 14 drinks/week for females or 21 drinks/week for males (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of Screening.
6. Treatment with an investigational drug within 30 days (or as determined by the local requirement) or 5 half lives preceding the first dose of study medication, whichever is longer.
7. Screening supine blood pressure ≥140 mm Hg (systolic) or ≥ 90 mm Hg (diastolic), following at least 5 minutes of supine rest. If blood pressure (BP) is ≥ 140 mm Hg (systolic) or 90 mm Hg (diastolic), the BP should be repeated two more times, following 2 minutes rest and the average of the three BP values should be used to determine the subject's eligibility.
8. Screening supine12 lead ECG demonstrating QTcf >450 or a QRS interval >120 msec. If QTcf exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated two more times and the average of the three QTc or QRS values should be used to determine the subject's eligibility.
9. Subjects with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study specific laboratory and confirmed by a single repeat, if deemed necessary:

   * Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transminase (SGOT) or alanine aminotransferase (ALT)/serum glutamic pyruvic transminase (SGPT) 1.5x upper limit of normal (ULN);
   * Total bilirubin 1.5 x ULN; subjects with a history of Gilbert's syndrome may have a direct bilirubin measured and would be eligible for this study provided the direct bilirubin is ULN.
10. Male subjects with partners currently pregnant; male subjects able to father children who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for at least 28 days after the last dose of investigational product or longer based upon the compound's half life characteristics.
11. For Part 1 and Part 3 specific: Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose of study medication. As an exception, acetaminophen/paracetamol may be used at doses of ≤ 1 g/day. Limited use of non prescription medications that are not believed to affect subject safety or the overall results of the study may be permitted on a case by case basis following approval by the sponsor.
12. For Part 2 specific: Systemic therapy with any of the following cytochrome P450 (CYP) 3A4 strong and moderate inhibitors/inducers within 7 days or 5 half lives (whichever was longer) prior to the first dose of study medication, or during the study: phenobarbital, carbamazepine, phenytoin, rifampin, rifabutin, St. John's Wort, bosentan, modafinil, nafcillin, aprepitant, ciprofloxacin, boceprevir, clarithromycin, conivaptan, grapefruit juice, itraconazole, ketoconazole, mibefradil, nefazodone, posaconazole, telaprevir, telithromycin, voriconazole, aprepitant, diltiazem, erythromycin, fluconazole, verapamil and human immunodeficiency virus (HIV) protease inhibitors (eg, indinavir, ritonavir, nelfinavir, atazanavir, amprenavir, fosamprenavir, etc).
13. For Part 2 specific: sensitive CYP3A substrates or CYP3A substrates with narrow therapeutic index within 7 days or 5 half lives (whichever was longer) prior to the first dose of study medication, or during the study. However, this exclusion may be removed if the Part 1 results suggest low risk.
14. Herbal supplements and hormone replacement therapy must be discontinued 28 days prior to the first dose of study medication.
15. Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 56 days prior to dosing.
16. History of sensitivity to heparin or heparin induced thrombocytopenia.
17. Unwilling or unable to comply with the Lifestyle Guidelines described in this protocol.
18. Subjects who are investigational site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the Investigator, or subjects who are Pfizer employees directly involved in the conduct of the study.
19. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
20. For Cohorts 3 5 in Part 1 specific: Subjects with a history of significant active bleeding, coagulation disorder or clinically significant finding on PT/PTT/INR at Screening.
21. For Cohorts 3 5 in Part 1 specific: Subjects with lower spinal malformations (on physical examination or lumber X ray), local spinal/skin infection, or other abnormalities that would exclude puncture (LP).
22. For Cohorts 3 5 in Part 1 specific: Subjects with allergy to lidocaine or its derivative.
23. Use of tobacco or nicotine containing products in excess of the equivalent of 5 cigarettes per day.
24. Subjects who answer "Yes" to the Columbia Suicide Severity Rating Scale (C SSRS) questions 4 or 5. In addition, subjects deemed by the investigator to be at significant risk of suicidal or violent behavior should be excluded.
25. Subjects who have attempted suicide in the past.
26. Subjects who have unexplained history of sudden death in their family.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Maximum Observed PF-06648671 Plasma Concentration (Cmax) | 0-24 hours on day 1 and 7 and 0-72 hours on day 14
  Cmax on day 1, 7 and day 14 in part 1, Cmax on day 1 and 14 in part 2
PF-06648671 Plasma Area Under the Curve from Time Zero to 24 hour after dosing (AUC24) | 0-24 hours on day 1 and 7 and 0-72 hours on day 14
  AUC24 on day 1, 7 and 14 in part 1, day 1 and 14 in part 2
Time to Reach Maximum Observed Plasma concentration (Tmax) | 0-24 hours on day 1 and 7 and 0-72 hours on day 14
  Tmax on day 1, 7 and 14 in part 1, day 1 and 14 in part 2
Plasma Decay half life | 0-24 hours on day 1 and 7 and 0-72 hours on day 14
  t1/2 post last dose on Day 14
Oral clearance (CL/F) | 0-24 hours on day 1 and 7 and 0-72 hours on day 14
  CL/F on day 14
Volume of distribution (Vz/F) | 0-24 hours on day 1 and 7 and 0-72 hours on day 14
  Vz/F on day 14
Observed PF-06648671 CSF concentration | 0 hr on day 1 and 0 hr on day 14 or 15
  PF-06648671 CSF concentration on day 1 and day 14 (cohort 3) or day 15 (cohorts 5, 6 and 8) prior to dosing in part 1
Accumulation factor of AUC24 | 0-24 hours on day 1 and 7 and 0-72 hours on day 14
  accumulation of PF-06648671 plasma AUC24 on day 7 and day 14 relative to day 1 in part 1, AUC on day 14 relative to day 1 in part 2
Accumulation factor of Cmax | 0-24 hours on day 1 and 7 and 0-72 hours on day 14
  PF-06648671 plasma Cmax on day 7 and 14 relative to day 1 in part 1, day 14 to day 1 in part 2
% parent drug in urine (Ae%) | 0-24 hr on day 14
  percentage of parent drug recovered in urine over 24 hours on day 14 in part 1 and part 2
Renal clearance (CLr) | 0-24 hours on day 14
  Renal clearance of PF-06648671 on day 14
CSF Abeta 40 and 42 concentration change from baseline | 0 hr on day 1 and 0 hr on day 14 or 15
  CSF Abeta 40 and 42 concentration on day 14 (cohort 3) or on day 15 (cohorts 5, 6 and 8) prior to dosing compared to day 1 baseline
Plasma AUC of midazolam alone vs co-administration with PF-06648671 in optional part 3 | 0-24hr on day 1 and 0-48hr on day 14
  the AUC ratio of midazolam between day 14 in period 2 vs day 1 in period 1 in optional part 3
Plasma Cmax of midazolam alone vs co-administration with PF-06648671 in optional part 3 | 0-24hr on day 1 and 0-48hr on day 14
  the Cmax ratio of midazolam between day 14 in period 2 vs day 1 in period 1 in optional part 3

SECONDARY OUTCOMES:
CSF Abeta 37, 38 and total concentration change from baseline | 0 hr on day 1 and 0 hr on day 14
  if possible, CSF abeta 37, 38 and total concentration on day 14 prior to dosing compared to day 1 prior to dosing in cohort 3 to 5 in part 1 only
Plasma Abeta change from baseline | 0-24hr on day 1 and 0-72hr on day 14
  Plasma abeta 40 and 42 and total abeta concentration change from baseline at multiple timepoints

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium

REFERENCES:
- [Derived] Ahn JE, Carrieri C, Dela Cruz F, Fullerton T, Hajos-Korcsok E, He P, Kantaridis C, Leurent C, Liu R, Mancuso J, Mendes da Costa L, Qiu R. Pharmacokinetic and Pharmacodynamic Effects of a gamma-Secretase Modulator, PF-06648671, on CSF Amyloid-beta Peptides in Randomized Phase I Studies. Clin Pharmacol Ther. 2020 Jan;107(1):211-220. doi: 10.1002/cpt.1570. Epub 2019 Sep 11. PMID 31314925
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7991002&StudyName=An%20Investigator-and-subject%20Blind%2C%20Phase%201%20Study%20To%20Characterize%20The%20Safety%2C%20Tolerability%2C%20Pharmacokinetics%2C%20And%20Pharmacodynamics%20Of%20Repeat%20Doses%20Of%20Pf-06648671%20In%20Healthy%20Adult%20Subjects%20And%20Healthy%20Elderly%20Subjects